CLINICAL TRIAL: NCT04545580
Title: A Randomized, Placebo-controlled, Double-blind, Parallel-group, Multi-center, Proof-of-concept Study to Assess the Efficacy and Safety of BAY 1817080 in Patients With Overactive Bladder (OAB) Over a 12-week Treatment Period
Brief Title: Clinical Study to Evaluate the Treatment Effect and Safety of BAY1817080 in Patients With Overactive Bladder (OAB)
Acronym: OVADER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19733; 2019-002575-34 (EudraCT Number)
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Overactive Bladder
Keywords: Urinary Bladder, Overactive; OAB; Urinary incontinence; Urinary urgency; Urgency; Micturition
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment period: Placebo (Placebo Comparator): This arm consists of participants who complete the run-in period, and are still eligible, according to all in- and exclusion criteria for diagnosis of OAB with UUI based on bladder diary baseline data. Participants will be randomized to 12 weeks of double-blind treatment with matching placebo.
  Interventions: Drug: Placebo
- Treatment period: BAY1817080 (Experimental): This arm consists of participants who complete the run-in period, and are still eligible, according to all in- and exclusion criteria for diagnosis of OAB with UUI based on bladder diary baseline data. Participants will be randomized to 12 weeks of double-blind treatment with BAY1817080.
  Interventions: Drug: BAY1817080

INTERVENTIONS:
Drug: Placebo — Matching placebo for BAY1817080, will be taken twice daily orally as tablet(s)
  Arms: Treatment period: Placebo
Drug: BAY1817080 — BAY1817080 will be taken twice daily orally as tablet(s)
  Arms: Treatment period: BAY1817080

SUMMARY:
The aim of the study is to determine how well the drug BAY1817080 works in OAB patients with urgency urinary incontinence (UUI), defined as involuntary leakage of urine, accompanied or immediately preceded by a sudden compelling desire to void.

BAY1817080 is a new drug under development which blocks proteins expressed on the sensory nerves in the bladder. These nerves seem to overreact in OAB patients.

This study will test if the treatment with BAY1817080 will reduce the frequency of OAB symptoms. The frequency of OAB symptoms before the treatment and the frequency after 4, 8 and 12 weeks of treatment will be compared.

Another important objective of this study will be the assessment of BAY1817080 safety and tolerability in this patient population.

BAY1817080 will be compared to a "placebo". A placebo tablet looks like the study drug but does not have any medicine in it. Using a placebo helps to learn if the study drug works. Each participant is expected to take part in the study for about 5 months (around 20-22 weeks).

ELIGIBILITY:
Inclusion Criteria:

at screening：

* Adults ≥ 18 years of age at the time of signing the informed consent
* Have "wet" OAB symptoms (urgency, frequency and urinary incontinence) for ≥ 3 months prior to screening visit
* Women of childbearing potential (WOCBP) must agree to use acceptable effective or highly effective contraceptive methods
* Capable of giving signed informed consent
* Willing and able to complete the electronic bladder diary and questionnaires

at baseline (to be checked at V3, prior to randomization):

* Completion of all 3 days of 3-day electronic bladder diary during run-in phase
* Compliance of ≥80% with intake of study intervention during run-in
* Frequency of micturition on average ≥ 8 episodes/24 hours during the run-in phase according to 3-day electronic bladder diary
* Frequency of urgency urinary incontinence on average ≥ 1 episode/24 hours during the run-in phase according to 3-day electronic bladder diary

Exclusion Criteria:

* Polyuria known or based on the clinical evidence during the run-in phase recorded in the 3-day electronic bladder diary and the investigator´s clinical judgement
* Significant stress incontinence or mixed stress/urgency incontinence
* Post-void residual volume (PVR) > 150 mL at Visit 1 or at Visit 3
* In need of catheterization (indwelling or intermittent)
* Clinically significant urinary outflow obstruction
* Previous pelvic radiation, or previous or current malignant disease of pelvic organs
* Neurogenic bladder
* Bladder pain syndrome/interstitial cystitis
* Recurrent and/or symptomatic bladder stones
* Current symptomatic or recent (within 30 days prior to Visit 1), or recurrent (2 or more infections within 6 months, or > 3 infections within 12 months) urinary tract infection
* Unexplained macro- or micro-hematuria
* Diabetes insipidus
* Diabetes mellitus with inadequate glycemic control as indicated by HbA1C result of > 8% at screening
* Clinically significant cardiovascular or cerebrovascular disease
* Systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg
* Clinically significant abnormal electrocardiogram (ECG) at screening
* Moderate-to-severe hepatic impairment defined as Child-Pugh Class B or C
* Laboratory values outside the inclusion range (as specified in the laboratory manual and in the reports from the central laboratory) before start of study intervention, and considered clinically relevant
* At screening:

  * ALT above 2xULN OR
  * AST above 2xULN OR
  * total bilirubin greater than ULN OR
  * AP above 2x ULN OR
  * INR greater than ULN (unless on vitamin K antagonist treatment) OR
  * Positive hepatitis B virus surface antigen (HBsAg) OR
  * Positive hepatitis C virus antibodies (anti-HCV) and detection of mRNA (HCV-mRNA, only tested if hepatitis C virus antibodies were detected)
* Severe renal impairment as defined by estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2 calculated by Modification of Diet in Renal Disease (MDRD) formula
* Any other diseases or conditions that according to the investigator can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study intervention (e.g., excessively low body weight, Chronic bowel disease, Crohn's disease and ulcerative colitis)
* Any severe or unstable diseases or medical conditions including psychiatric disorders that might interfere with the conduct of the study, or could jeopardize the safety of the participant, or the interpretation of the results
* History of major depression within 2 years prior to screening, or a history of other major psychiatric disorder at any time (e.g., schizophrenia, bipolar disorder)
* Concurrent malignancy or history of cancer (except for adequately treated basal cell or squamous cell carcinoma of the skin) within the last 5 years prior to screening
* Intake of prohibited medication due to potential drug-drug interaction Use of other treatments that might interfere with the conduct of the study or the interpretation of the results e.g.

  * a) use of any drug treatment after start of study intervention intended for the OAB/UI symptoms other than the study intervention
  * b) neuromodulation therapy and intravesical treatment - less than 12 months prior to screening or at any time during the study
  * c) use of any treatment intended for other conditions but which can affect urinary bladder function during the study
  * d) Non-drug treatment (e.g. physical treatment or acupuncture): permitted only if initiated ≥4 weeks prior to Screening and planned to be continued during the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Average change from baseline over Week 4, 8 and 12 (end of treatment [EoT]) in mean number of urgency urinary incontinence (UUI) episodes/24 hours based on electronic bladder diary | From baseline up to 12 weeks

SECONDARY OUTCOMES:
Change from baseline to Week 12 (EoT) based on electronic bladder diary in mean number of UUI episodes/24 hours | From baseline up to 12 weeks
Change from baseline to Week 12 (EoT) based on electronic bladder diary in mean number of urinary incontinence (UI) episodes/24 hours | From baseline up to 12 weeks
Change from baseline to Week 12 (EoT) based on electronic bladder diary in mean number of micturition episodes/24 hours | From baseline up to 12 weeks
Change from baseline to Week 12 (EoT) based on electronic bladder diary in mean number of urgency episodes (Grade 3 or 4)/24 hours | From baseline up to 12 weeks
Change from baseline to Week 12 (EoT) based on electronic bladder diary in mean number of nocturia episodes/24 hours | From baseline up to 12 weeks
Change from baseline to Week 12 (EoT) based on electronic bladder diary in mean volume voided per micturition | From baseline up to 12 weeks
Incidence of adverse events | From the start of study intervention (at start of run-in) until the follow-up visit (up to 18 weeks)

CONTACTS AND LOCATIONS:
Locations (28):
- Australia (2):
  - Emeritus Research, Botany, New South Wales
  - Emeritus Research, Camberwell, Victoria
- Austria (2):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universität Innsbruck, Innsbruck
- Czechia (7):
  - Afimed s.r.o, Benešov
  - Gynekologie Cheb s.r.o., Cheb
  - G-Centrum Olomouc s.r.o. Dr. Skrivanek, Olomouc
  - GynCare MUDr. Michael Svec s.r.o., Pilsen
  - Urocentrum Praha, s.r.o., Prague
  - Androgeos - private center of urology and andrology, Prague
  - Fakultní nemocnice Bulovka, Prague
- Germany (4):
  - Urologicum Duisburg - Praxis Walsum, Duisburg, North Rhine-Westphalia
  - Überörtliche Gemeinschaftspraxis "Urologie Neandertal", Mettmann, North Rhine-Westphalia
  - Urologicum, Eisleben Lutherstadt, Saxony-Anhalt
  - Praxis Hr. Dr. M. Markov, Halle, Saxony-Anhalt
- New Zealand (2):
  - Canterbury Urology Research Trust, Christchurch
  - Tauranga Urology Research Limited, Tauranga
- Poland (5):
  - Medico Praktyka Lekarska, Krakow
  - NZOZ NOVITA, Specjalistyczne Gabinety Lekarskie S.C, Lublin
  - Centrum Urologiczne Sp. z o.o., Mysłowice
  - NZOZ Heureka, Piaseczno
  - Przychodnia Lekarska Eskulap, Skierniewice
- Portugal (3):
  - CHULN - Hospital Santa Maria, Lisbon
  - Centro Hospitalar Universitario do Porto, Porto
  - CHUSJ - Hospital Sao Joao, Porto
- KK Women's and Children's Hospital, Singapore, Singapore
- Sweden (2):
  - Göteborgs Urologmottagning, Gothenburg
  - Urogyn, Solna

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Fletcher MC. Selectivity of the P2X3 receptor antagonist Eliapixant, and its potential use in the treatment of endometriosis. Purinergic Signal. 2022 Mar;18(1):1-3. doi: 10.1007/s11302-021-09831-5. Epub 2022 Jan 3. No abstract available. PMID 34978027
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field — http://clinicaltrials.bayer.com/